CLINICAL TRIAL: NCT00072267
Title: A Phase II Study of UCN-01 in Combination With Topotecan in Patients With Advanced Ovarian Cancer
Brief Title: UCN-01 and Topotecan in Treating Patients With Recurrent, Persistent, or Progressive Advanced Ovarian Epithelial, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-019; CDR0000339563 (Registry Identifier: PDQ (Physician Data Query)); NCI-6402
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; primary peritoneal cavity cancer; fallopian tube cancer; stage III ovarian epithelial cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — 7-hydroxystaurosporine; Topotecan

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, work in different ways to stop tumor cells from dividing so they stop growing or die. UCN-01 may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining UCN-01 with topotecan may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining UCN-01 with topotecan in treating patients who have recurrent, persistent, or progressive advanced ovarian epithelial, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of UCN-01 and topotecan, in terms of complete and partial objective response rates, in patients with recurrent, persistent, or progressive advanced ovarian epithelial, primary peritoneal, or fallopian tube cancer.

Secondary

* Determine the antitumor activity of this regimen, in terms of stable disease rates and duration of response, in these patients.
* Determine the progression-free, median, and overall survival of patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the relationship between clinical and pharmacodynamic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive UCN-01 IV over 3 hours on day 1 and topotecan IV over 30 minutes on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 19-33 patients will be accrued for this study within 5-11 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed ovarian epithelial, primary peritoneal, or fallopian tube cancer

  * Progressive, persistent, or recurrent disease
* Measurable disease outside prior radiotherapy field unless disease progression occurred after radiotherapy
* Tumor lesions accessible for biopsy

  * Patients with a medical contraindication to tumor biopsy may be allowed at the discretion of the principal investigator
* No more than 2 prior chemotherapy regimens

  * At least 1 regimen must have contained a platinum agent (i.e., carboplatin or cisplatin)
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal

* Creatinine no greater than ULN OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* No history of coronary artery disease
* No symptomatic cardiac dysfunction
* No cardiac pathology by electrocardiogram* NOTE: *Patients with symptomatic coronary artery disease must undergo an electrocardiogram

Pulmonary

* No symptomatic pulmonary dysfunction

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 8 weeks after study participation
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to UCN-01 or other study agents
* No insulin-dependent diabetes mellitus

  * Diabetes controlled by diet or oral hypoglycemic agents allowed at the discretion of the investigator
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior biologic therapy and recovered

Chemotherapy

* See Disease Characterisitcs
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior topotecan
* No other prior topoisomerase I inhibitors

Endocrine therapy

* More than 4 weeks since prior hormonal therapy and recovered

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 40% of bone marrow
* No prior mediastinal irradiation

Surgery

* More than 4 weeks since prior surgery and recovered

Other

* No other concurrent anticancer therapy
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hal W. Hirte, MD, FRCP(C), Principal Investigator — Margaret and Charles Juravinski Cancer Centre
Locations (4):
- Canada (4):
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario